CLINICAL TRIAL: NCT01203228
Title: Dose-reduced Versus Standard Conditioning Followed by Allogeneic Stem Cell Transplantation in Patients With MDS or sAML: A Randomised Phase III Study (RICMAC)
Brief Title: Dose-reduced Versus Standard Conditioning in MDS/sAML
Acronym: RICMAC
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: European Society for Blood and Marrow Transplantation (Network)
Collaborators: Pierre Fabre Medicament (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2005-002011-24; EBMT 42205525; NCT00682396 (obsolete NCT alias)
Record Dates: First submitted 2010-09-15; First posted 2010-09-16 (Estimated); Last update posted 2015-04-03 (Estimated); Status verified 2015-04

CONDITIONS: Myelodysplastic Syndromes; Secondary Acute Myeloid Leukemia
Keywords: Reduced Intensity conditioning; Myeloablative conditionig; Allogeneic stem cell transplantation; MUD
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — Busulfan; fludarabine phosphate; Bone Marrow Purging; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator): Myeloablative conditioning
  Interventions: Other: Myeloablative conditioning
- B (Experimental): Reduced Intensity Conditioning
  Interventions: Other: Reduced Intensity Conditioning

INTERVENTIONS:
Other: Reduced Intensity Conditioning — Busilvex®:
  6.4 mg/kg IBW i. v. day -7: 0.8 mg/kg IBW x 4 (2 hour infusion every 6 hours) day -6: 0.8 mg/kg IBW x 4 (2 hour infusion every 6 hours)
  or (if i.v.-application is not available)
  Busulfan:
  8.0 mg/kg BW p. o.: day -7: 4.0 mg/kg BW day -6: 4.0 mg/kg BW
  plus:
  Fludarabine:
  5 x 30 mg/m² BS i. v.: day -7: 30 mg/m² BS day -6: 30 mg/m² BS day -5: 30 mg/m² BS day -4: 30 mg/m² BS day -3: 30 mg/m² BS
  Other Names: Myleran; Sulphabutin; Busulphan; Leucosulfan; Myeloleukon; Citosulfan; Mielevcin; Milecitan; Fludara; Beneflur; Fludura; FAMP; 2-Fluoro-ara-AMP
  Arms: B
Other: Myeloablative conditioning — Busilvex®:
  12.8 mg/kg IBW i. v.; day -9: 0.8 mg/kg IBW x 4 (2 hour infusion every 6 hours) day -8: 0.8 mg/kg IBW x 4 (2 hour infusion every 6 hours) day -7: 0.8 mg/kg IBW x 4 (2 hour infusion every 6 hours) day -6: 0.8 mg/kg IBW x 4 (2 hour infusion every 6 hours)
  or (if i.v.-application is not available):
  Busulfan:
  16.0 mg/kg BW p. o.; day -9: 4.0 mg/kg BW day -8: 4.0 mg/kg BW day -7: 4.0 mg/kg BW day -6: 4.0 mg/kg BW
  plus:
  Cyclophosphamide:
  120 mg/kg BW i. v.; day -4: 60 mg/kg BW day -3: 60 mg/kg BW
  Other Names: Myleran; Sulphabutin; Busulphan; Leucosulfan; Myeloleukon; Citosulfan; Mielevcin; Milecitan; cyclophosphamide; Procytox; Cytoxan; Cyclophosphan; Cytophosphan; Claphene; Cyclostin; Endoxan
  Arms: A

SUMMARY:
In this trial dose reduced conditioning is compared to standard conditioning followed by allogeneic stem cell transplantation from related or unrelated donors in patients with MDS or secondary AML.

Conditioning is the very high dose chemotherapy treatment that is given in the days before the stem cell transplant.

The hypothesis is that a dose reduced conditioning will reduce the non-relapse mortality from 40% to 20% at one year after allogeneic stem cell transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Disease: Cytologically proven primary or therapy-related myelodysplastic syndrome (MDS), either as

  * refractory anaemia (RA) according FAB or RA with or without dysplasia according WHO,
  * refractory anaemia with ringsideroblasts (RARS) according FAB or RARS with or without dysplasia according WHO,
  * refractory anaemia with excess of blasts (RAEB) according FAB or RAEB I or RAEB II according WHO,
  * refractory anaemia with excess of blast in transformation (RAEB T) according FAB,
  * CMML (dysplastic type) according WHO,
* or secondary acute myeloid leukaemia (sAML).
* Blast count < 20 percent in bone marrow with or without chemotherapy at time of transplantation.
* Patient eligible for standard and dose-reduced conditioning as per local guideline.
* Patient age 18 - 60 years if donor is a HLA-matched unrelated donor (HLA-A, HLA-B, HLA-DRB1 and HLA-DQB1) (one mismatch allowed):
* Patient age 18 - 65 years if donor is a HLA-matched related donor ((HLA-A, HLA-B, HLA-DRB1 and HLA-DQB1) (one anti¬gen-mismatch allowed):
* No major organ dysfunction.
* Written informed consent of the patient.

Exclusion Criteria:

* Blasts > 20 % in bone marrow at time of transplantation
* No written informed consent.
* Central nervous involvement.
* Severe irreversible renal, hepatic, pulmonary or cardiac disease, such as
* Total bilirubin, SGPT or SGOT > 2 times upper the normal level.
* Left ventricular ejection fraction < 30 %.
* Creatinine clearance < 30 ml/min.
* DLCO < 35 % and/or receiving supplementary continuous oxygen.
* Positive serology for HIV.
* Pregnant or lactating women.
* Patients with a life-expectancy of less than six months because of another debilitating disease.
* Serious psychiatric or psychological disorders.
* Invasive fungal infection at time of registration.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2004-05; Primary Completion 2015-01 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
non-relapse mortality | every 6 months for safety and in the final analysis at one year after allogeneic stem cell transplantation

SECONDARY OUTCOMES:
organ related toxicity of conditioning | every 6 months for safety and in the final analysis at day +30 after allogeneic stem cell transplantation
Incidence of aGVHD | every 6 months for safety and in the final analysis at day +100 after allogeneic stem cell transplantation
incidence of cGVHD | every 6 months for safety and in the final analysis at one year after allogeneic stem cell transplantation
overall survival | every 6 months for safety and in the final analysis at 2 years after allogeneic stem cell transplantation
event-free survival | every 6 months for safety and in the final analysis at 2 years after allogeneic stem cell transplantation
cumulative incidence of relapse | every 6 months for safety and in the final analysis at 2 years after allogeneic stem cell transplantation
VOD | every 6 months for safety and in the final analysis at day +100 after allogeneic stem cell transplantation
infection incidence | every 6 months for safety and in the final analysis at day +100, 1 year and 2 years after allogeneic stem cell transplantation
Haematopoeitic recovery | every 6 months for safety and in the final analysis at day +30 after allogeneic stem cell transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Nicolaus Kröger, MD, Study Chair — Universitätsklinikum Hamburg-Eppendorf; Axel R Zander, MD, Principal Investigator — University Hospital Hamburg-Eppendorf, Germany; Ghulam J Mufti, MD, Principal Investigator — King's College Hospital London, United Kingdom; Marie Robin, MD, Principal Investigator — Hopital Saint-Louis Paris, France; Kathrin Haifa Al-Ali, MD, Principal Investigator — University Hospital Leipzig, Germany; Dietger Niederwieser, MD, Principal Investigator — University Hospital Leipzig, Germany; Giorgio Lambertenghi Deliliers, Principal Investigator — IRCCS Ospedale Maggiore of Milan, Italy; Domink Heim, Prof., Principal Investigator — University Hospital, Basel, Switzerland; Liisa Volin, MD, Principal Investigator — Helsinki University Central Hospital, Finland; Stefano Guidi, MD, Principal Investigator — Careggi Hospital - Florence, Italy; Augustin Ferrant, MD, Principal Investigator — Cliniques Universitaires St. Luc Bruxelles, Belgium; Afanasyer Boris, Principal Investigator — SPB Pavlov Medical Univ, St. Petersburg, Russia; Kai Hubel, Principal Investigator — University of Cologne; Peter Dreger, Principal Investigator — Univ Hospital Heidelberg - Germany; Martin Gramatzlle, Principal Investigator — University Hospital Münster - Germany; Gerhard Behre, Principal Investigator — Martin-Luther-Universitaet Halle-Wittenberg - Germany; Martin Gramatzlle, Principal Investigator — Univ Hospital Kiel - Germany; Allione Bernardino, Principal Investigator — Santi Antonio E Biagio
Locations (14):
- Germany (9):
  - University Hospital, Cologne
  - University Hospital, Düsseldorf
  - Martin-Luther-Universität Halle-Wittenberg, Halle
  - University Hospital Eppendorf, Hamburg
  - University Hospital, Heidelberg
  - UKSH Campus Kiel, Kiel
  - University Hospital, Leipzig
  - Universitätsklinikum Munster, Münster
  - University Hospital, Tübingen
- Italy (3):
  - Santi Antonio e Biagio, Alessandria
  - Ospedale di Careggi, Florence
  - Ospedale Maggiore di Milano, Milan
- Radboud University MC, Nijmegen, Netherlands
- SPb State I. Pavlov Medical University, Saint Petersburg, Russia

REFERENCES:
- See also: Related Info — http://www.ebmt.org/Contents/Pages/Default.aspx